CLINICAL TRIAL: NCT06209606
Title: Treatment of Patients with Relapsed/Refractory Multiple Myeloma with Ruxolitinib, Methylprednisolone and Lenalidomide: Using Changes in Serum B-Cell Maturation Antigen (BCMA) or International Multiple Working Group (IMWG) Criteria to Determine Disease Progression in Order to Add Lenalidomide to Those Failing the Ruxolitinib/Methylprednisolone Combination
Brief Title: Pilot Study Using Changes in Serum BCMA to Determine Disease Progression in Multiple Myeloma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I-RUX-20-52
Record Dates: First submitted 2024-01-08; First posted 2024-01-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ruxolitinib; Lenalidomide; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; methyl prednisolonate

STUDY DESIGN:
Intervention Model Description: This is a pilot, multicenter, open-label study evaluating the utility of using increases in serum BCMA > 25% versus IMWG criteria to determine disease progression among patients with RRMM treated with ruxolitinib and methylprednisolone to determine when to add lenalidomide to the regimen. Subjects that were treated with ruxolitinib with methylprednisolone and showed disease progression will have lenalidomide added to their regimen. PD is defined by either change in sBCMA (≥ 25% increase from nadir) or by standard IMWG criteria, whichever occurs first. PD will be confirmed by two consecutive tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rux + Steroid (Experimental): Subject will receive Ruxolitinib Oral Tablet [Jakafi] at 15mg BID, and Methylprednisolone at 40mg QOD until disease progression. Lenalidomide at 10mg QD will be added to the treatment (Ruxolitinib, Methylprednisolone) once disease progression was confirmed.
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Methylprednisolone
- Rux + Steroid + Len (Experimental): Ruxolitinib Oral Tablet [Jakafi] at 5mg, 10mg or 15mg BID, Lenalidomide Oral at 5mg or 10mg QD and Methylprednisolone Oral at 40mg QOD. (Dose varies during dose escalation portion of the study)
  Interventions: Drug: Ruxolitinib Oral Tablet [Jakafi]; Drug: Lenalidomide; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet [Jakafi] — Ruxolitinib will be administered on days 1-28 of the treatment cycle.
  Other Names: Ruxolitinib, Jakafi
Drug: Lenalidomide — Lenalidomide will be administered on Days 1-21 of the treatment cycle.
  Other Names: Revlimid
  Arms: Rux + Steroid + Len
Drug: Methylprednisolone — Methyl-prednisolone will be administered on Days 1-28 of the treatment cycle.
  Other Names: Depo-Medrol, Solu-Medrol, Methyl Prednisolonate

SUMMARY:
This is a phase 1, multicenter, open-label study evaluating the safety and efficacy of ruxolitinib, steroids and lenalidomide among MM patients who currently show progressive disease using BCMA to test progression.

DETAILED DESCRIPTION:
In recent years, new and more effective drugs have become available for the treatment of multiple myeloma (MM), resulting in a dramatic increase in median overall survival (OS).1 Therapeutic options have expanded to include immune-based approaches such as daratumumab and elotuzumab.2 The clinical course of MM is highly variable, and relapsing/refractory (RR)MM more so, with periods of response followed by periods of relapse. Improvements in predicting and determining individual patient outcome would allow for more effective and timely treatment interventions.

Over the last several years, we have identified a new serum biomarker, B cell maturation antigen (BCMA), for monitoring patients with MM. Changes in serum (s)BCMA quickly identify changes in the clinical status of MM and it is also a promising new prognostic marker. Specifically, we demonstrated that compared to healthy donors, patients with MM showed elevated levels of sBCMA.3 These levels were positively correlated with the proportion of plasma cells in bone marrow biopsies and changes in monoclonal (M)-protein and serum free light chain (SFLC) levels and indicated a patient's current clinical status.3 Importantly, sBCMA levels were also independent of renal function and maintained independent significance when tested against other known prognostic markers for MM including age, serum β-2-microglobulin, hemoglobin, and presence of bone disease. Furthermore, we demonstrated that increases in sBCMA by > 25% from start of any new therapy predicted a markedly shorter progression free survival (PFS) and occurred much more quickly than those observed with standard biomarkers to monitor the course of MM including M-protein and SFLC levels.

To further validate sBCMA as a disease status biomarker for MM, we have incorporated monitoring of sBCMA for all patients participating in several ongoing clinical trials. Specifically, patients participating in a Phase 1 study of ruxolitinib, methylprednisolone and lenalidomide for RRMM patients, were monitored weekly for sBCMA and standard MM markers during their first treatment cycle and monthly thereafter. We determined the safety and efficacy of this novel, all oral combination consisting of the Janus kinase 1/2 inhibitor ruxolitinib in combination with lenalidomide and methylprednisolone.5 Successive cohorts of participants (3 participants per cohort) were given the following doses of drugs, all oral (PO): Dose Level 0: ruxolitinib 5 mg twice a day (BID), methylprednisolone 40 mg every other day (QOD) and lenalidomide 5 mg daily (QD) on days 1-21 of a 28-day cycle; Dose Level 1: ruxolitinib 10 mg BID, methylprednisolone 40 mg QOD, and lenalidomide 5 mg QD on days 1 21 of a 28-day cycle; Dose Level 2: ruxolitinib 15 mg BID, methylprednisolone 40 mg QOD, and lenalidomide 5 mg QD on days 1 21 of a 28-day cycle), and Dose Level 3: ruxolitinib 15 mg BID, methylprednisolone 40 mg QOD and lenalidomide 10 mg QD on days 1 21 of a 28-day cycle. Dose Level 3 was the maximum administered dose.

Data analysis on the first 28 patients treated with this triple combination demonstrated promising safety and efficacy profiles.5 Specifically, the clinical benefit rate (CBR) and overall response rate (ORR)7 were 46% and 38%, respectively.5 No dose-limiting toxicities occurred. Grade 3 or grade 4 adverse events (AEs) included anemia (18%), thrombocytopenia (14%), and lymphopenia (14%). Most common serious AEs (SAE) included sepsis (11%) and pneumonia (11%). Notably, all 12 responding patients were refractory to lenalidomide and steroids.

To date, we have enrolled a total of 49 patients. Forty are evaluable for safety and efficacy.8 The CBR and ORR were 47% and 37%, respectively. Responses included 1 complete response (CR), 4 very good partial responses (VGPR), 10 partial responses (PR), and 4 minimal responses (MR), and 16 and 5 patient showed stable disease (SD) and progressive disease (PD), respectively. Notably, all 19 patients achieving > MR were refractory to lenalidomide (i.e., progressed while on or within 8 weeks of receiving the last dosage of this drug). PFS for all evaluable patients was 4.0 months with the median follow-up time of 3.0 months (range, 0.2 13.3). The median follow-up time for the responding patients was 5.4 months (0.9 13.3) with the duration of response (DOR) of 5.0 months. This all oral regimen was well tolerated, and reversible Grade 3/4 cytopenias occurred in only a small minority of patients.

We analyzed sBCMA levels for these patients and demonstrated that its baseline levels predicted PFS and increases of > 25% occurred more rapidly than those observed with M protein or SFLC and predicted for a much shorter PFS.9 Specifically, serum BCMA was a faster predictor than International Myeloma Working Group (IMWG) criteria of disease progression for 67% of the MM patients showing disease progression, and no patient showed progression more rapidly using IMWG criteria than sBCMA.

Furthermore, an expansion of the ongoing Phase 1 study is evaluating the combination of ruxolitinib 15 mg BID and methylprednisolone 40 mg QOD continuously without lenalidomide in this same patient population. Subjects are enrolled and treated with this two-drug combination until disease progression. Twenty-nine patients were enrolled in the doublet combination, and the ORR and CBR were both 45% (2 VGPR, 11 PR, 0 MR). Per study design, once disease progression occurred as determined using IMWG criteria, lenalidomide at 10 mg PO daily on days 1 21 of a 28-day cycle was added to the regimen. To date, 19 subjects have been enrolled in this portion of the study and 17 patients have completed at least 2 full cycles of lenalidomide-containing therapy. Ten patients have responded (3 PR and 7 MR) while 4 patients exhibited SD and 5 patients had PD.

These results show that the combination of ruxolitinib and steroids is active for treating RRMM and that the addition of lenalidomide upon disease progression will overcome disease progression in many patients. These results provide the basis for the current trial which will use monitoring of sBCMA levels and IMWG criteria to more quickly allow addition of lenalidomide to patients failing the two-drug combination.

Therefore, in this pilot study involving patients with RRMM initially treated with ruxolitinib and methylprednisolone, we specifically propose to use changes in sBCMA levels (> 25% increase from its nadir level) or conventional indicators of disease progression per IMWG criteria (changes in M-protein and SFLC levels), whichever occurs first, to determine when to add lenalidomide to patients failing the doublet combination of ruxolitinib and methylprednisolone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria to be eligible to enroll in this study.

  1. Has a diagnosis of MM based on standard criteria as follows:

     Major criteria:

  <!-- -->

  1. Plasmacytomas on tissue biopsy
  2. BM plasmacytosis (greater than 30% plasma cells)
  3. Monoclonal immunoglobulin spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL or kappa or lambda light chain excretion greater than 1 g/day on 24-hour urine protein electrophoresis

     Minor criteria:

  <!-- -->

  1. BM plasmacytosis (10% to 30% plasma cells)
  2. Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
  3. Lytic bone lesions
  4. Normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL

Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:

* any 2 of the major criteria
* major criterion 1 plus minor criterion 2, 3, or 4
* major criterion 3 plus minor criterion 1 or 3
* minor criteria 1, 2, and 3, or 1, 2, and 4

  2. Currently has MM with measurable disease, defined as:
* a monoclonal immunoglobulin spike on serum electrophoresis of at least 0.5 g/dL and/or urine monoclonal protein levels of at least 200 mg/24 hours
* for patients without measurable serum and urine M-protein levels, an involved SFLC > 100 mg/L or abnormal SFLC ratio
* for patients with IgD MM, a monoclonal immunoglobulin IgD of at least 5500 mg/L or meet other measurable disease eligibility criteria

  3. Currently has progressive MM and has received at least 2 prior regimens including lenalidomide, a proteasome inhibitor, and an anti-CD38 antibody:
* Patients are considered relapsed when they progress greater than 8 weeks from their last dose of treatment
* Patients are refractory when they progress while currently receiving the treatment or within 8 weeks of its last dose

  4. Ruxolitinib naïve

  5. Understand and voluntarily sign an informed consent form before receiving any study-related procedure that is not part of normal medical care, with the understanding that consent may be withdrawn at any time without prejudice to their future medical care

  6. Able to adhere to the study visit schedule and other protocol requirements

  7. ECOG performance status of ≤ 2 at study entry

  8. Life-expectancy of greater than 3 months

  9. Laboratory test results within these ranges at Screening and confirmed at enrollment prior to drug dosing on Cycle 1, Day 1:
* Absolute neutrophil count ≥ 1.5 x 109/L

  o If the bone marrow is extensively infiltrated (≥ 70% plasma cells) then ≥ 1.0 x 109/L
* Platelet count ≥ 75 x 109/L

  o Patients must not have received platelet transfusion for at least 7 days prior to receiving screening platelet count
  * If the bone marrow is extensively infiltrated (≥ 70% plasma cells) then ≥ 50 x 109/L
  * If patient have creatinine clearance of less than 60mL/min, patient's platelet count must be greater than 150 x 109/L
* Hemoglobin ≥ 8.0 g/dL within 21 days prior to enrollment

  o Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion must have been at least 7 days prior to obtaining screening hemoglobin.
* Calculated or measured CrCl > 60 mL/minute per Cockcroft-Gault (Appendix 3)
* Total bilirubin levels ≤ 2.0 mg/dL
* AST (SGOT) and ALT (SGPT) ≤ 2 x ULN
* Serum potassium 3.0 - 5.5 mEq/L

  10. Patients receiving lenalidomide (Part 2 of the study) must be registered into the mandatory REVLIMID REMS™ program, and be willing and able to comply with the requirements of the REVLIMID REMS™ program

  11. FCBP† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting ruxolitinib + methylprednisolone and must either commit to continued abstinence from heterosexual intercourse or use acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, and at least 28 days before she starts taking ruxolitinib with or without lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.

  †A FCBP (female of childbearing potential) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; and 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

  12. Able to take antiplatelet therapy if platelet count is above 30 x 109/L. Options include aspirin (acetylsalicylic acid, ASA) at 81 or 325 mg/daily and warfarin or low molecular weight heparin if ASA-intolerant

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are not to be enrolled in the study:

  1. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
  2. Plasma cell leukemia (> 2.0 × 109/L circulating plasma cells by standard differential)
  3. Primary amyloidosis
  4. Non-hematologic malignancy within the past 5 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
  5. Patients with uncontrolled infections
  6. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

     * Myocardial infarction within 6 months prior to enrollment
     * New York Heart Association (NYHA) Class II or greater heart failure or uncontrolled angina
     * Clinically significant pericardial disease
     * Severe uncontrolled ventricular arrhythmias
     * Echocardiogram or MUGA evidence of LVEF below institutional normal within 28 days prior to enrollment
     * Electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening must be documented by the investigator as not medically relevant.
     * Severe hypercalcemia, i.e., serum calcium ≥ 12 mg/dL (3.0 mmol/L) corrected for albumin
  7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
  8. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
  9. Undergone major surgery within 28 days prior enrollment or has not recovered from side effects of such therapy (vertebroplasty or kyphoplasty is not considered to be a major surgery; however, the investigator is to discuss enrollment of a subject with a recent history of kyphoplasty with the medical monitor).
  10. Pregnant or breastfeeding females (lactating females must agree not to breast feed while taking lenalidomide)
  11. Received the following prior therapy:

      * Chemotherapy within 3 weeks of study drugs
      * Corticosteroids (>20 mg/daily prednisone or equivalent) within 3 weeks of study drugs to ensure that steroid dose intensity at the beginning of the treatment is not altered by administration of steroids prior to the study. Consumption of steroids within 3 weeks of the treatment may interfere with efficacy and side effects due to differences of steroid intensity.
      * Immunotherapy, antibody therapy, immunomodulatory drugs, or proteasome inhibitors within 3 weeks of study drugs
      * Extensive radiation therapy within 28 days before study drugs. Receipt of localized radiation therapy does not preclude enrollment.
      * Use of any other experimental drug or therapy within 28 days of study drugs
      * JAK inhibitor including ruxolitinib
  12. Strong CYP3A4 inhibitors, strong CYP3A4 inducers and fluconazole doses >200 mg daily within 5 half-lives before study drugs. (For example, clarithromycin has half-life of 4 hours so washout period for clarithromycin is 20 hours.)
  13. Known hypersensitivity to compounds of similar chemical or biological composition to thalidomide and lenalidomide or steroids.
  14. Concurrent use of other anti-cancer agents or treatments
  15. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
  16. Known positivity for human immunodeficiency virus (HIV), hepatitis B or C, and /or active tuberculosis (TB) including subjects with latent TB or with the risk factor for activation of latent TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression (TTP) | 54 months
  * To establish the utility of using an increase in sBCMA levels > 25% or IMWG criteria for disease progression to direct this therapeutic approach, TTP will be measured, where TTP is defined as a number of days between the start of treatment (cycle 1 day 1) and PD. PD is defined by either change in sBCMA (≥25% increase from its nadir levels) or by standard IMWG criteria (using sM-protein and SFLC assessments), whichever occurs first. PD will be confirmed by two consecutive tests.
  * Duration of response 1 (DOR1), defined as the time from the first response to progressive disease as determined by either changes in sBCMA or IMWG criteria (whichever occurs first) while patients are on ruxolitinib and methylprednisolone treatment
  * Duration of response 2 (DOR2), defined as the time from the first response to progressive disease as determined by standard IMWG criteria while patients on ruxolitinib, lenalidomide and methylprednisolone treatment

SECONDARY OUTCOMES:
Safety and Tolerability | 54 months
  • Occurrence of adverse events throughout the study, graded via Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 criteria
Efficacy and Overall Response | 54 months
  * Efficacy of treatment will be assessed by the overall response rate (ORR; ORR = CR + VGPR + PR) and clinical benefit rate (CBR; CBR = CR + VGPR + PR + MR) of the doublet and triplet combinations
  * PFS1 as defined based on the length of time that patient was receiving therapy consisting of ruxolitinib with steroids until PD or death from any cause as determined by either an increase in sBCMA of ≥25% from its nadir or using IMWG criteria
  * PFS2 as defined based on the length of time that patient was receiving ruxolitinib, lenalidomide and steroid therapy to the time they reached disease progression as determined by the standard IMWG criteria or death from any cause
  * PFS from start of study treatment to disease progression as determined by the standard IMWG criteria or death from any cause including receiving treatment with ruxolitinib, lenalidomide and steroid

CONTACTS AND LOCATIONS:
Overall Officials: James Berenson, MD, Principal Investigator — Oncotherapeutics
Locations (1):
- Berenson Cancer Center, West Hollywood, California, United States